CLINICAL TRIAL: NCT03681860
Title: Open Label, Dose Escalation and Age De-escalation for ChAdOx1 85A in Ugandan Adults and Adolescents, Followed by a Phase IIa Randomised, Open-label Trial Among Adolescents Comparing ChAdOx1 85A Prime Followed by MVA 85A Boost Versus BCG Re-vaccination.
Brief Title: EMaBS TB Vaccine Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB042
Record Dates: First submitted 2018-09-04; First posted 2018-09-24 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Safety; Immunogenicity
Keywords: BCG; Tuberculosis; Vaccination
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Masking Description: This will be an open label trial as it will not be possible to blind either volunteers or clinic staff to the allocation. However, laboratory staff will be blinded to the allocation of the volunteers as they undertake the immunological assays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 Dose Escalation Adults (Other): 3 adults who are parents of EMaBS participants, to receive ChAdOx1 85A at 5 x10^9 vp
  Interventions: Biological: ChAdOx185A
- Group 2 Dose Escalation Adults (Other): 3 adults who are parents of EMaBS participants, to receive ChAdOx1 85A at 2.5 x10^10 vp
  Interventions: Biological: ChAdOx185A
- Group 3 Age De-escalation Adolescents (Other): 3 adolescents who are EMaBS participants, to receive ChAdOx1 85A at 5 x10^9 vp
  Interventions: Biological: ChAdOx185A
- Group 4 Age De-escalation Adolescents (Other): 3 adolescents who are EMaBS participants, to receive ChAdOx1 85A at 2.5 x10^10 vp
  Interventions: Biological: ChAdOx185A
- Group 5/6 Randomised Comparison (Experimental): 30 adolescents who are EMaBS participants, to receive ChAdOx1 85A at 2.5 x10^10 vp followed by MVA85A boost versus 30 adolescents who are EMaBS participants, to receive BCG revaccination
  Interventions: Biological: ChAdOx185A; Biological: MVA85A; Biological: BCG

INTERVENTIONS:
Biological: ChAdOx185A — ChAdOx1 85A is an adenoviral vaccine based on a vector that is a chimpanzee adenovirus isolate Y25 expressing the M.tb antigen 85A. Adenoviruses are attractive candidates for use as viral vectors and have been used as vaccine vectors for a number of conditions; however, the use has been limited by the high level of anti-vector immunity present in humans in whom adenovirus is a ubiquitous infection. This has led to the consideration of simian adenoviruses, which are not known to cause pathology or illness in humans and to which the prevalence of anti-vector antibodies is low. The ChAdOx1 vector has been developed by the University of Oxford and been used with different inserts for vaccination, for example the vaccine ChAdOx1 NP+M1 has demonstrated an excellent safety profile in the Influenza trial FLU004. A BCG - ChAdOx1 85A - MVA85A prime boost regime is more protective than BCG alone in mice.
Biological: MVA85A — Modified vaccinia virus Ankara (MVA) is a highly-attenuated strain of vaccinia virus which cannot replicate in human cells. It is known to be highly immunogenic in UK adults but has been less immunogenic in African children and infants. It is suitable for use as a viral vector in a prime-boost regime in new vaccine development. It has an excellent safety record as it was administered intradermally to approximately 120,000 people during the smallpox eradication campaign, and has since been used in numerous clinical trials of candidate vaccines against viral, mycobacterial and protozoal infections.
  Arms: Group 5/6 Randomised Comparison
Biological: BCG — BCG is the only vaccine currently approved for use against Tuberculosis.
  Arms: Group 5/6 Randomised Comparison

SUMMARY:
The study will commence with a dose-escalation and age de-escalation study in healthy adults and adolescents from the previous Entebbe Mother and Baby Study (EMaBS) in Entebbe, Uganda, focusing on ChAdOx1 85A, to provide safety data for ChAdOx1 85A in this population. These measures are not required for MVA85A since this vaccine has been more widely used, including among adolescents in Uganda, and the dose has been standardised. ChAdOx1 85A dose escalation and age de-escalation will be followed by a Phase IIa randomised trial comparing the immunogenicity of ChAdOx1 85A and MVA85A with the immunogenicity of BCG revaccination. ChAdOx1 85A and MVA85A will be administered via the intramuscular route. The target dose for the Phase IIa trial is 2.5x10^10 viral particles (vp) because the lower dose is expected to have lower immunogenicity, based on the Oxford study, TB034. Data from the Oxford study suggest that this dose will be well tolerated. However, if this dose is not tolerated then the lower dose will be used. The dose of MVA85A will be 1 x 10^8 plaque-forming units (pfu) in the groups in which it is given. There will be 6 study groups with 3 to 30 volunteers in each group.

Dose escalation for ChAdOx1 85A in adults Group 1:

The first three adults will receive ChAdOx1 85A at 5 x10^9 vp.

Group 2:

The next three adults will be enrolled after safety data has been reviewed by the trial management team to one week after ChAdOx1 85A vaccination in group 1. These adults will receive ChAdOx1 85A at 2.5 x10^10 vp.

Age de-escalation and dose escalation for ChAdOx1 85A in adolescents Group 3:

The first three adolescents will be enrolled after safety data has been reviewed to one week after ChAdOx1 85A vaccination in group 2. These three adolescents will receive ChAdOx1 85A at 5 x10^9 vp Group 4. The next three adolescents will be enrolled after safety data has been reviewed to one week after ChAdOx1 85A vaccination in group 2. These three adolescents will receive ChAdOx1 85A at 2.5 x10^10 vp.

Randomised comparison of ChAdOx1 85A-MVA85A versus BCG revaccination:

Once safety data has been reviewed for groups 1 to 4 to one week post ChAdOx1 85A vaccination, recruitment to the randomised trial will commence. Sixty adolescents will be randomised, 30 (group 5) to receive ChAdOx1 85A at 2.5 x10^10 vp followed by MVA85A boost and 30 (group 6) to receive BCG revaccination.

BCG will be obtained from the Serum Institute of India, an approved provider for Uganda, and used at the standard dose of 0.1mL. BCG will be given intradermally.

DETAILED DESCRIPTION:
This trial will be financed by a research grant from Medical Research Council. The reference number of the grant held by MRC-UKRI is MC_UU_00027/5.

ELIGIBILITY:
Inclusion Criteria:

* Resident within the study area and planning to be resident in the study area for the duration of the study or participants with documented good attendance who are willing to attend as required
* Participant in the Entebbe Mother and Baby Study; healthy; aged 12 to 17 [or, for adults, a parent or guardian of a participant; healthy; aged 18 to 49]
* Documented immunisation within two weeks of birth with BCG Russia (BCG-I strain from Moscow, Serum Institute of India, India) [adolescents only]
* BCG scar or documented previous BCG immunisation [adults only]
* No relevant findings in medical history or on physical examination
* Written informed consent by parent or guardian [or by the volunteer themselves, for adults]
* Written informed assent by subject [for adolescents]
* Agreed to refrain from blood donation during the trial [adults only; adolescents under age 18 are not eligible to give blood]
* Agree to avoid pregnancy for the duration of the trial (female only)
* Able and willing (in the Investigator's opinion) to comply with all the study requirements

Exclusion Criteria:

* Clinical, radiological, or laboratory evidence of current active TB disease
* Laboratory evidence at screening of latent M.tb infection as indicated by a positive ELISPOT response to ESAT6 or CFP10 antigens
* Previous treatment for active or latent tuberculosis infection
* Shared a residence with an individual who has started on anti-tuberculosis treatment, or been diagnosed with culture or smear-positive pulmonary tuberculosis, within six months prior to day 0
* Received a TST within 90 days prior to day 0
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer, cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness, drug or alcohol abuse
* History of serious psychiatric condition or disorder
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents within 2 months prior to enrollment
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the study vaccine, including eggs
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the volunteer in the study
* Positive HBsAg, HCV or HIV antibodies
* Use of an investigational medicinal product or non-registered drug, live vaccine, or medical device other than the study vaccine for 30 days prior to dosing with the study vaccine, or planned use during the study period
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
* Female currently lactating, confirmed pregnancy or intention to become pregnant during the trial period
* Screening blood sample positive for malaria by microscopy

Ages: 12 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Safety: Solicited Adverse Events | 30 months
  Actively and passively collected data on adverse events
Immunogenicity: T-cell response to 85A | 30 months
  T-cell Interferon-gamma ELIspot response to antigen 85A

SECONDARY OUTCOMES:
Immunogenicity: antibodies to 85A | 30 months
  ELISA antigen 85A to show antibody response to antigen 85A in blood/serum after vaccination
Exploratory immunology: Flow cytometry | 30 months
  Innate and B-cell flow cytometry panel to characterize surface cell markers on B-cells and Neutrophils after vaccination
Exploratory immunology: gene expression | 30 months
  Gene expression array (CHIP) to identify the genes expressed during immune response to vaccination
Exploratory immunology: mycobacterial killing assay | 30 months
  Assay to show ability or improvement of immune cells to kill mycobacteria after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Professor, Principal Investigator — University of Oxford
Locations (2):
- MRC/UVRI and LSHTM Uganda Research Unit, Entebbe Hospital, Entebbe, Uganda
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT03681860/Prot_SAP_001.pdf